CLINICAL TRIAL: NCT01376661
Title: Outcome Assessment of an Active Surveillance Program for Low Risk Prostate Cancer: An Observational Study
Status: Terminated | Type: Observational
Why Stopped: Early termination due to PI's decision to discontinue research activities.
Sponsor: St. Joseph Hospital of Orange (Other)
Responsible Party: Sponsor
Other Study IDs: 09-009 Active Surveillance
Record Dates: First submitted 2011-06-03; First posted 2011-06-20 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Active Surveillance; Low risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active Surveillance/ Prostate Cancer

SUMMARY:
The purpose of this research study is to monitor the feasibility and outcome of the Active Surveillance Program for men with low risk prostate cancer.

DETAILED DESCRIPTION:
The purpose of this observational study is to prospectively monitor the outcome associated with men who meet the eligibility criteria for low risk prostate cancer and elected to participate in the active surveillance program at The Center for Cancer Prevention and Treatment at St. Joseph Hospital. We hope to demonstrate that men who are compliant with a closely monitored active surveillance program for low risk prostate cancer will achieve favorable outcomes by: 1) avoiding the side effects of definitive therapy that may not be necessary; 2) retaining quality of life (QOL) and normal activities; 3) avoiding unnecessary treatment; and 4) decreased health care costs. In addition, we will monitor the possible adverse outcomes that may be associated with the active surveillance program including suboptimal response and/or greater side effects due to delayed initiation of therapy; psychological impact on the patients and caregivers due to anxiety of living with an untreated cancer and/or the requirement for frequent medical examination and periodic prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histological documented adenocarcinoma of the prostate either newly diagnosed or previously diagnosed. Subjects who are diagnosed more than 3 months prior to time of enrollment in the active surveillance program must have biopsy repeated.
* PSA < 10 ng/ml within 1 month of program enrollment
* Clinical stage less than or equal to T2a
* Biopsy sampling with at least 10-12 cores
* Gleason score less than or equal to 3 + 3
* No more than 2 cores involved
* No core more than 50% involved
* Eligible for definitive therapy
* Able to provide informed consent
* Able to complete a QOL questionnaire
* Able to comply with the scheduled follow-up appointments

Exclusion Criteria:

* See inclusion criteria for eligibility

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with low risk prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of enrolled subjects who remain compliant free until disease progression. | 10 years
  This measurement will monitor the feasibility of the Active Surveillance Program for men with low risk prostate cancer

SECONDARY OUTCOMES:
Percentage of enrolled subjects who require definitive therapy | 10 years
Quality of Life as measured by patient survey. | 10 Years
Overall survival | 10 years
  This will be a measurement of the treatment outcome.
Cost/Benefit Analysis | 10 Years
  This measure will determine the feasibility of the Active Surveillance Program.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Greenberger, MD, Principal Investigator — St. Joseph Hospital of Orange
Locations (1):
- St. Joseph Hospital of Orange, Orange, California, United States